CLINICAL TRIAL: NCT04586309
Title: Improving the Mental Health of Resident Physicians and Fellows : Reducing Burnout & Enhancing Resilience Through Transcendental Meditation
Brief Title: Improving the Mental Health of Resident Physicians and Fellows Through Transcendental Meditation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Feasibility
Sponsor: University of Arizona (Other)
Collaborators: David Lynch Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2008969193
Record Dates: First submitted 2020-10-02; First posted 2020-10-14 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Burnout, Professional; Stress, Psychological; Depression; Job Stress
Keywords: transcendental meditation; resilience; burnout
MeSH Terms: conditions — Burnout, Professional; Stress, Psychological; Depression; Occupational Stress; Burnout, Psychological | interventions — Meditation

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to the TM training (group 1), or delayed TM training (group 2). Study outcomes will be assessed at baseline and at 1 and 3 months post-training. Participants who are assigned to group 2 , will receive the TM training following the three month assessment, and then complete assessments at 1 and 3 months post-training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early TM Training (Experimental): This group will receive training in Transcendental Meditation and will complete assessments at baseline, 1 month and 3 months.(3 assessments in total).
  Interventions: Behavioral: Transcendental meditation
- Delayed TM training (Active Comparator): This arm will complete the baseline, 1 month and 3 month assessments and then will receive the TM training, followed by additional 1 month and 3 month post-training assessments (5 in total)
  Interventions: Behavioral: Transcendental meditation

INTERVENTIONS:
Behavioral: Transcendental meditation — Instruction in the TM technique is taught over five sessions.
  1. Introductory session-Review of previous scientific research on the TM program and a vision of possible benefits; Preparation- discussion of the mechanics and origin of the TM technique After the introductory session, a Personal Interview is conducted telephonically-with a teacher of the TM program.
  2. Personal Instruction-individual one-on-one instruction in the TM technique. The student learns the mechanics of the TM technique. At the conclusion of this class the student is able to meditate properly.
  3. First Day of Verification of Correct Practice and Further Instruction.
  4. Second Day of Verification of Correct Practice-understanding the mechanics of the TM technique from personal experiences.
  5. Third Day of Verification of Correct Practice-understanding the mechanics of the development of higher human potential and wellness.

SUMMARY:
This proposal aims to optimize resident physician and fellow wellness and performance at Banner University Medical Center through an evidence-based stress reduction program, Transcendental Meditation (TM). It is particularly timely due to the enormous pressure and stress that residents face as front-line workers during the current 2019 novel coronavirus (COVID-19) pandemic.

Participants will be randomly assigned to the TM training (group 1), or delayed TM training (group 2). Study outcomes will be assessed at baseline and at 1 and 3 months post-training. Participants who are assigned to group 2 , will receive the TM training following the three month assessment, and then complete assessments at 1 and 3 months post-training.

These assessment tools look at anxiety (Generalized Anxiety Disorder Scale-GAD-7), depression (Patient Health Questionnaire (PHQ-9), insomnia (Pittsburgh Sleep Quality Index PSQI), psychological distress (Brief Symptom Inventory BSI18), burnout (Maslach Burnout Inventory-MBI), resilience (Conner-Davidson Resilience Scale- RISC), and alcohol use (Alcohol Use Disorder Identification Test - AUDIT).

DETAILED DESCRIPTION:
Up to one hundred resident and fellow physicians employed by Banner Health will participate in the project. Participants will be randomly assigned to either the TM program or to a delayed TM training, treatment-as-usual control group . Study outcomes will be assessed at baseline, 1-month and 3-month post-training , with change in burnout as the primary outcome. Control subjects (aka delayed TM training or Group 2) will be eligible to learn TM after completing 3 month post-testing. Group 2 will also complete post-training assessments at 1-month and 3-months post-training. The total duration of this project will be 60 months.

Two experienced certified TM instructors will conduct the instruction. All certified TM teachers have been extensively trained in the teaching of the TM program, including teaching the course of instruction, verifying continued correctness of effortless practice of the technique, and conducting additional follow-up sessions. The same standardized TM course sequence will be used for all study participants.

Outline of Transcendental Meditation Program: TM group will involve 10 total sessions over 12 weeks (about 75 minutes per session). The core instruction in the TM technique will involve a course of instruction, taught over five sessions. The five core instruction sessions will include:

1. Introductory session-Review of previous scientific research on the TM program and a vision of possible benefits; Preparation- discussion of the mechanics and origin of the TM technique(75 minutes- group session); After the introductory session, a Personal Interview is conducted telephonically-with a teacher of the TM program. The participant completes a brief interview form prior to the call. The interviewer (a teacher with the TM program) reviews the form with the participant.

   The four classes of TM instruction adhere to a standardized teaching protocol and are conducted by certified teachers of the Transcendental Meditation program trained and approved by the Transcendental Meditation organization.
2. Personal Instruction-individual one-on-one instruction in the TM technique (75 minutes). The student learns the mechanics of the TM technique. At the conclusion of this class the student is able to meditate properly.
3. First Day of Verification of Correct Practice and Further Instruction (90 minutes-group session); The first follow-up session provides information to help students incorporate TM into their daily life.
4. Second Day of Verification of Correct Practice-understanding the mechanics of the TM technique from personal experiences (90 minutes-group session); The second session provides information about how the meditation reduces stress and improves health
5. Third Day of Verification of Correct Practice-understanding the mechanics of the development of higher human potential and wellness (90 minutes-group session). The third session reviews students' experiences both during and after meditation, and provides further instruction to support their ongoing home practice.

Following the initial phase of the intervention (5 sessions), there will be 5 additional group sessions of 45-60minutes each provided once a month for the remainder of the 6-month intervention period. These sessions will include: a) discussion of personal experiences and verification of correctness of practice of the TM technique, and b) knowledge of the human potential and its relationship to mental and physical health.

Compliance with treatment sessions will be defined as attending at least 70% of the treatment sessions. Subjects randomized to the TM group will continue with their usual care.

No research data is collected during the sessions described above.

Although it is the intent for all of these sessions to be conducted at the Tucson Transcendental Meditation Center, in small physically distanced groups of participants wearing whatever level of personal protective equipment is being recommended by the CD at the time of the session, in the event that in person sessions are not possible, the group sessions will be held virtually through Zoom video conferencing. Additionally, participants may be able to complete sessions 3-5 over the TM App (a series of pre-recorded lectures).

For participants who choose to use the TM App, they will be asked to create an account through the app, and will be given the opportunity to review the Terms of Service and Privacy Policies. Maharishi Foundation International (the owners/developers of the App) monitor the participants progress through the digital content so that they know when to release the next session (as described above). Participants can also use the App to time their meditation sessions, although this is not required.

Home Practice: Home practice will consist of two 20-minute TM sessions daily - morning and evening. Compliance with TM practice will be defined as meditating at least once a day. Participants will complete a home practice questionnaire at 1 month and 3 months (attached as an addendum-will be included in the REDCap bundle with assessments).

Delayed TM training/Control Condition: Subjects randomized to the control group will continue with their usual care. Control subjects will be invited to learn the TM program after 3-month post-training assessment. If they chose to complete the TM training, they will be subject to the same training as Group 1, and the same assessments after the end of their training.

ELIGIBILITY:
Inclusion Criteria:

1. Full-time Resident physicians or Fellows employed by Banner Health
2. 18 years or older
3. Some participants included will have treated COVID-19 patients or be working at locations where COVID-19 patients are being treated.
4. Willing to take part in either group assignment (randomized to either immediate start or TM training, or delayed TM training)
5. Willing to complete baseline, 1-month and 3-month post- assessments
6. If being treated with psychoactive medications, the maintenance of a stable regimen for at least two months before enrollment (by self-report).

Exclusion Criteria:

1. Already instructed in the Transcendental Meditation technique
2. Currently unstable psychotic symptoms, mania or bipolar disorder as demonstrated by self-report, or psychiatric hospitalizations in the past six months;
3. Current suicidal or homicidal ideation with intent or plan.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Burnout | baseline
  Maslach Burnout Inventory- Participants respond to each prompt 0-6, high score in first 2 sections, low score in third may indicate risk of burnout.
Burnout | 1 month
  Maslach Burnout Inventory- Participants respond to each prompt 0-6, high score in first 2 sections, low score in third may indicate risk of burnout.
Burnout | 3 month
  Maslach Burnout Inventory- Participants respond to each prompt 0-6, high score in first 2 sections, low score in third may indicate risk of burnout.

SECONDARY OUTCOMES:
Resilience | baseline
  Connor-Davidson Resilience Scale- Participants respond to each prompt 0-5 x 25 items, low score indicates poor resilience.
Resilience | 1 month
  Connor-Davidson Resilience Scale- Participants respond to each prompt 0-5 x 25 items, low score indicates poor resilience.
Resilience | 3 months
  Connor-Davidson Resilience Scale- Participants respond to each prompt 0-5 x 25 items, low score indicates poor resilience.
Alcohol use | baseline
  AUDIT: Alcohol Use Disorders Identification Test- Participants respond to 10 items with 0-4, higher score more concerning for alcohol use disorder.
Alcohol use | 1 month
  AUDIT: Alcohol Use Disorders Identification Test- Participants respond to 10 items with 0-4, higher score more concerning for alcohol use disorder.
Alcohol use | 3 months
  AUDIT: Alcohol Use Disorders Identification Test- Participants respond to 10 items with 0-4, higher score more concerning for alcohol use disorder.
Depression | baseline
  PHQ-9: Patient Health Questionnaire- Participants answer each prompt (not all all, some days, most days, nearly every day) higher numbers indicate greater depressive symptoms.
Depression | 1 month
  PHQ-9: Patient Health Questionnaire- Participants answer each prompt (not all all, some days, most days, nearly every day) higher numbers indicate greater depressive symptoms.
Depression | 3 months
  PHQ-9: Patient Health Questionnaire- Participants answer each prompt (not all all, some days, most days, nearly every day) higher numbers indicate greater depressive symptoms.
Sleep Quality | baseline
  PSQI: Pittsburgh Sleep Quality Index- Participant answers 19 questions in 7 sections, Seven sections are combined for global score of 0-21 where ) is no problems and 21 is problems in all areas.
Sleep Quality | 1 month
  PSQI: Pittsburgh Sleep Quality Index- Participant answers 19 questions in 7 sections, Seven sections are combined for global score of 0-21 where ) is no problems and 21 is problems in all areas.
Sleep Quality | 3 months
  PSQI: Pittsburgh Sleep Quality Index- Participant answers 19 questions in 7 sections, Seven sections are combined for global score of 0-21 where ) is no problems and 21 is problems in all areas.
Distress | baseline
  BSI18: Brief Symptom Inventory 18- Participants answer 18 questions on 0-4 scale. Higher numbers indicate more distress.
Distress | 1 month
  BSI18: Brief Symptom Inventory 18
Distress | 3 months
  BSI18: Brief Symptom Inventory 18
Anxiety | baseline
  GAD7: Generalized Anxiety Disorder 7- Participants answer 7 questions 0-3. Higher scores indicate greater anxiety,
Anxiety | 1 month
  GAD7: Generalized Anxiety Disorder 7- Participants answer 7 questions 0-3. Higher scores indicate greater anxiety,
Anxiety | 3 months
  GAD7: Generalized Anxiety Disorder 7- Participants answer 7 questions 0-3. Higher scores indicate greater anxiety,

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lai J, Ma S, Wang Y, Cai Z, Hu J, Wei N, Wu J, Du H, Chen T, Li R, Tan H, Kang L, Yao L, Huang M, Wang H, Wang G, Liu Z, Hu S. Factors Associated With Mental Health Outcomes Among Health Care Workers Exposed to Coronavirus Disease 2019. JAMA Netw Open. 2020 Mar 2;3(3):e203976. doi: 10.1001/jamanetworkopen.2020.3976. PMID 32202646
- [Background] Valosek L, Link J, Mills P, Konrad A, Rainforth M, Nidich S. Effect of Meditation on Emotional Intelligence and Perceived Stress in the Workplace: A Randomized Controlled Study. Perm J. 2018;22:17-172. Published 2018 Oct 29. doi:10.7812/TPP/17-172
- See also: Information from David Lynch Foundation regarding grant — http://healthehealersnow.org
- See also: Information about transcendental meditation and other TM research — http://TM.org